CLINICAL TRIAL: NCT01393184
Title: Prospective, Randomized, Controlled, Phase II，Multiple Centered Clinical Trial of Nimotuzumab Combined With Radiotherapy for Senile Locally Advanced SCCHN
Brief Title: Safety and Efficacy Study of Target Therapy Combined With Radiotherapy to Treat Senile Locally Advanced SCCHN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University (Other)
Collaborators: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Peking University, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-IST-SCCHN-040
Record Dates: First submitted 2011-06-24; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-03

CONDITIONS: SCCHN
Keywords: Target therapy
MeSH Terms: interventions — nimotuzumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy + Nimotuzumab (Experimental): 1. Radiotherapy (RT) Technique: IMRT, Rapid Arc, Tomotherapy Total dose: GTV 70 Gy & CTV 60 Gy/33F
  2. Nimotuzumab (Nimo) weekly Nimo (200 mg) × 8, started 1 w before RT
  Interventions: Drug: Nimotuzumab and Radiotherapy
- Radiotherapy (RT) (Active Comparator): Radiotherapy (RT) Technique: IMRT, Rapid Arc, Tomotherapy Total dose: GTV 70 Gy & CTV 60 Gy/33F
  Interventions: Drug: Nimotuzumab and Radiotherapy

INTERVENTIONS:
Drug: Nimotuzumab and Radiotherapy — Nimotuzumab (Nimo)： Nimotuzumab weekly Nimo (200 mg) × 8, started 1 w before RT
  Other Names: Nimotuzumab combined with radiotherapy

SUMMARY:
Radiotherapy alone is generally the only treatment in old patients with SCCHN. No evidence indicates combination with EGFR Target therapy can bring benefit for the patients. Senile Society is coming in China, the mean age in Beijing reaches 80 years old. A valuable treatment with efficacy and safety is needed for senile patient with SCCHN. The purpose of the study "Prospective, Randomized, Controlled, Phase II Multiple Centered Clinical Trial of Nimotuzumab Combined with Radiotherapy for Senile Locally Advanced SCCHN" was sponsored to evaluate the efficacy and safety for Nimotuzumab Combined with Radiotherapy in Senile SCCHN patients.

DETAILED DESCRIPTION:
condition: Senile Locally Advanced SCCHN. Intervention: Drug:Nimotuzumab. Arm A: Radiotherapy+Nimotuzumab; Arm B: Radiotherapy alone. Phase: Phase 2

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form
* Age 65-85，both genders
* HNSCC Confirmed by pathology
* Primary site of oral cavity, oropharynx, hypopharynx, larynx
* Stage Ⅲ/ⅣA,B
* Primary lesions can be measured
* Karnofsky's Performance Scale ≥60
* Life expectancy of more than 6 months
* Haemoglobin≥100g/L ,WBC ≥3.5×109/L, platelet count≥90×109/L
* Hepatic function: ALT、AST< 1.5 x ULN, TBIL< 1.5 x ULN
* Renal function: Creatinine < 1.5 x ULN

Exclusion Criteria:

* Received other anti EGFR monoclonal antibody treatment
* Previous chemotherapy or radiotherapy
* Participation in other interventional clinical trials within 1 month
* Other malignant tumor (except of non-melanoma skin Cancer or carcinoma in situ of cervix)
* History of serious allergic or allergy
* History of Serious lung or heart disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate: complete response + partial response on RECIST evaluation system | 1-month after treatment
Evaluate the Safety of Nimotuzumab Combined with Radiotherapy for old patients. Record the Number and Grade of Participants with Adverse Events as a Measure of Safety and Tolerability | participants will be followed during the treatment,an expected average of 6 weeks
Objective response rate: complete response + partial response on RECIST | 3-months after treatment

SECONDARY OUTCOMES:
Evaluate the Local control Rate in 2 years. | up to 2 years
Evaluate the Quality of Life（QoL）of Senile Locally Advanced SCCHN treated by Nimotuzumab Combined with Radiotherapy or Radiotherapy alone. | participants will be followed during the treatment,an expected average of 6 weeks
  Record the subjective description of the patients by themself according to the QOL table.
Evaluate the overall survival of the patient in 2 years. | up to 2 years
Evaluate the progression free survival of the patient in 2 years. | up to 2 years
Evaluate the Quality of Life（QoL）of Senile Locally Advanced SCCHN treated by Nimotuzumab Combined with Radiotherapy or Radiotherapy alone. | every 3 months after treatment
  Record the subjective description of the patients by themself according to the QOL table.
Evaluate the Local control Rate in 3 years. | up to 3 years
Evaluate the Local control Rate in 5 years. | up to 5 years
Evaluate the overall survival of the patient in 3 years. | up to 3 years
Evaluate the overall survival of the patient in 5 years. | up to 5 years
Evaluate the progression free survival of the patient in 3 years. | up to 3 years
Evaluate the progression free survival of the patient in 5 years. | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sun Yan, MD, Principal Investigator — Peking University, School of Oncology, Beijing Cancer Hospital & Institute